CLINICAL TRIAL: NCT04300946
Title: Effects of the Magnetic Transcranial Stimulation (TMS) in Healthy Volunteers
Brief Title: Time Prediction and Cerebellum: Magnetic Transcranial Stimulation (TMS) in Healthy Volunteers
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7650
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- TMS on the cerebellum followed by placebo TMS: TMS preceding the time prediction and language tests
  Interventions: Device: TMS targeted on the cerebellum
- Placebo TMS followed by TMS on the cerebellum: TMS preceding the time prediction and language tests
  Interventions: Device: TMS targeted on the cerebellum
- TMS on the cerebellum set in time on waiting periods
  Interventions: Device: TMS targeted on the cerebellum
- TMS on the cerebellum not set in time on waiting periods
  Interventions: Device: TMS targeted on the cerebellum

INTERVENTIONS:
Device: TMS targeted on the cerebellum — Impact on EEG performance (preparation wave in temporal tasks) of cerebellar stimulation by MSD in healthy subjects. The contrast between the post-stimulation effects of verrum stimulation and placebo stimulation will indicate the magnitude of the effect and will allow us to optimize the type of protocol that may be useful in schizophrenia.

SUMMARY:
The aim of the study is to check the role of the cerebellum in time prediction in healthy volunteers, by means of magnetic transcranial stimulation targeted on the cerebellum, and recording of behavioural measures indexing time prediction

ELIGIBILITY:
Inclusion Criteria:

* Participant, male or female, between 18 and 60 years old
* Subject affiliated to a social health insurance scheme (beneficiary or entitled person)
* Subject who has dated and signed an informed consent form
* For a woman of childbearing age, negative pregnancy test and effective contraception throughout the study

Exclusion Criteria:

* - Participant with substance use disorders (as defined by DSM-V)
* Participants taking benzodiazepines and related substances (in the period before inclusion, for a duration equivalent to 5 half-lives of the product), cannabis (in the 2 months before inclusion) or hallucinogenic substances (in the period before inclusion, for a duration equivalent to 5 half-lives of the product).
* Participant with neurological pathology or sequelae
* Participant with Attention Deficit Hyperactivity Disorder (ADHD)
* Participant with a borderline personality disorder
* Participant with disabling sensory impairments, including visual acuity (corrected, if applicable) < 0.8 (due to use of visual material) (Freiburg Vision Test, Bach 1996)
* Participant deprived of liberty or subject to the safeguard of justice
* Participant under guardianship or curatorship
* Participant in a period of exclusion defined by another clinical study or participant in a study that may impact on research results
* Pregnant or breastfeeding woman
* Subject with a contraindication to performing an MRI or TMS: presence of non-removable ferromagnetic body, prosthesis, pacemaker, medication delivered by an implanted pump, vascular clip or stent, heart valve or ventricular lead, certain intracerebral clips, cochlear implants, history of epilepsy, skin pathology at the point of contact with the electrodes.
* Subject with a history of major neurological or psychiatric illness with current psychotropic medication (i.e., antidepressant, thyroid regulator, antipsychotic, benzodiazepine and related drugs, or hypnotic).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
EEG index of time expectation | 40 minutes
  CNV
EEG index of time expectation | 40 minutes
  beta oscillation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Strasbourg, Strasbourg, France